CLINICAL TRIAL: NCT02106962
Title: The Use of Topical Tranexamic Acid and Bacitracin in Dialysis Patients
Brief Title: Use of Topical Tranexamic Acid and Bacitracin in Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: California Institute of Renal Research (Other)
Collaborators: Imprimis Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Boiskin, MD, California Institute of Renal Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001-Boiskin
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Arteriovenous Fistula
Keywords: hemodialysis; fistula; clotting; tranexamic acid; bacitracin
MeSH Terms: conditions — Arteriovenous Fistula; Fistula; Thrombosis | interventions — Tranexamic Acid; Bacitracin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clotting time Using Tranexamic Acid 5% (Experimental): Measure Native AV Fistula clotting time after dialysis using 5% Tranexamic Acid compared to normal Clotting time of Native AV Fistula after dialysis
  Interventions: Drug: Topical Tranexamic Acid 5% with bacitracin
- Clotting Time Using Tranexamic Acid 25% (Experimental): Measure Native AV Fistula clotting time after dialysis using 25% Tranxemic Acid compared to normal clotting time of native AV Fistula after dialysis
  Interventions: Other: Topical Tranexamic Acid 25% with bacitracin

INTERVENTIONS:
Drug: Topical Tranexamic Acid 5% with bacitracin — Selected participants received a fixed amount of tranexamic acid 5 %and bacitracin applied with compression up to 3 times (13 minutes total) per hemodialysis fistula needle site.
  Other Names: Cyklokapron
  Arms: Clotting time Using Tranexamic Acid 5%
Other: Topical Tranexamic Acid 25% with bacitracin — Selected participants received a fixed amount of tranexamic acid 25%and bacitracin applied with compression up to 3 times (13 minutes total) per hemodialysis fistula needle site.
  Other Names: Cyklokapron
  Arms: Clotting Time Using Tranexamic Acid 25%

SUMMARY:
This study will investigate how the use of Tranexamic acid and Bacitracin applied to the bleeding site after the hemodialysis fistula needle is removed will affect Time to Clot and Infection Rate

DETAILED DESCRIPTION:
Visit 1 - Initial Application:

* A patient candidate identified by the PI who meets all of the inclusion criteria and none of the exclusion criteria will be consented for the study.
* The medical history will be collected from the subject.
* The subject will receive routine hemodialysis
* Directly after the completion of hemodialysis, the following study drug application steps will occur:

  1. Site 1 Initial Compression: Apply fixed amount of Tranexamic acid and bacitracin 5% or 25% to gauze and compress for 3 minutes to needle site 1.
  2. Site 2 Initial Compression: Apply fixed amount of Tranexamic acid and bacitracin 5% or 25% to gauze and compress for 3 minutes to needle site 2.
  3. Second Compression per site: If bleeding has not stopped, repeat application with new gauze and same amount of ointment to each respective site and compress for 5 minutes more at each site.
  4. Third Compression per site: If after the second application and compression the bleeding persists repeat both application and compression for another 5 minutes (total time would be 13 minutes at this step).
  5. Test Failure: If after the third application to each needle site there is still bleeding, the testing would be considered a failure and routine procedures should be utilized to stop the bleeding.
* Any adverse events will be collected.

Visit 2 - Follow-Up:

• The 1 week follow up visit will be performed to review study drug application site and to collect any adverse events reported by subject

The clotting time will be compared to the clotting time at a different dialysis session in which no treatment will be used

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients with fistulas (native arterio-venous)

Exclusion Criteria:

* Previous sensitivity to or adverse reaction to Tranexamic acid or Bacitracin.
* Active infection.
* Stenosis of fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Boiskin, MD, Principal Investigator — California Institute of Renal Research
Locations (3):
- United States (3):
  - Fresenius Medical Care - Kearny Mesa, San Diego, California
  - California Insitute of Renal Research, San Diego, California
  - Fresenious Medical Care - Rancho, San Diego, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Tranexamic Acid 5%: Topical Tranexamic Acid 5% with bacitracin applied to the arterio-venous fistula site after completing dialysis, to measure clotting time.
- Topical Tranexamic Acid 25%: Topical Tranexamic Acid 25% with bacitracin applied to the arterio-venous fistula site after completing dialysis, to measure clotting time.
Period: Overall Study
Arm/Group | Topical Tranexamic Acid 5% | Topical Tranexamic Acid 25%
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: dialysis subjects using arteriovenous fistula for dialysis access
Groups:
- Topical Tranexamic Acid and Bacitracin 5%: Topical Tranexamic Acid 5% with bacitracin applied to the arterio-venous fistula site after completing dialysis, to measure clotting time in the same participants that did not receive treatment at a subsequent dialysis session
- Tranexamic Acid and Bacitracin 25%: Topical Tranexamic Acid 25% with bacitracin applied to the arterio-venous fistula site after completing dialysis, to measure clotting time in the same participants that received treatment but at a subsequent dialysis session.
- Total: Total of all reporting groups
Arm/Group | Topical Tranexamic Acid and Bacitracin 5% | Tranexamic Acid and Bacitracin 25% | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Clotting TIme
Description: After completing dialysis, the clotting time of the arteriovenous fistula of each participant was measured, using either Tranexamic Acid 5% or Tranexamic Acid 25% and compared to the regular clotting time of the AV Fistula without using the Tranexamic Acid
Time Frame: 13 minutes
Measure: Mean (Full Range); unit: minutes
Arm/Group | Clotting Time Using Tranexamic Acid 5% | Clotting Time Using Tranexamic Acid 25%
Number analyzed (Participants) | 9 | 8
minutes | 6 [3 to 15] | 8 [3 to 15]

2. Secondary Outcome: Local Infection
Description: After using Tranexamic Acid and Bacitracin, local infection rate measured at the end of study
Time Frame: 2 months
Population: no local infection in any particioant
Measure: Mean (Full Range); unit: participants
Groups:
- Topical Tranexamic Acid 5%: Measure clotting time of Native arteriovenous fistula after applying topical Tranexamic Acid 5% compared with normal clotting time
- Topical Tranexamic Acid 25 %: Measure clotting time of Native arteriovenous fistula using Tranexamic acid 25% compared with normal clotting time
Arm/Group | Topical Tranexamic Acid 5% | Topical Tranexamic Acid 25 %
Number analyzed (Participants) | 8 | 9
participants | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Groups:
- Topical Tranexamic Acid 5% and Bacitracin: Topical Tranexamic Acid 5% with bacitracin applied to the arterio-venous fistula site after completing dialysis, to measure clotting time.
- Topical Tranexamic Acid 25% and Bacitracin: Topical Tranexamic Acid 25% with bacitracin was applied to the arterio-venous fistula site after completing dialysis, to measure clotting time at a subsequent dialysis session.
Arm/Group | Topical Tranexamic Acid 5% and Bacitracin | Topical Tranexamic Acid 25% and Bacitracin
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No